CLINICAL TRIAL: NCT05379686
Title: Low-Dose Glucagon and Advanced Hybrid Closed-Loop System for Prevention of Exercise-Induced Hypoglycaemia in People With Type 1 Diabetes
Brief Title: Glucagon and Advanced HCL System to Prevent Exercise-Induced Hypoglycaemia in People With Type 1 Diabetes
Acronym: HYPOAVOID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 85256; 2021-004993-68 (EudraCT Number)
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 Diabetes; Hypoglycemia; Exercise; Glucagon; Hybrid closed-loop system
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity | interventions — Glucagon-Like Peptide 1; Glucagon

STUDY DESIGN:
Intervention Model Description: Two-arm open-label intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150 ug glucagon before exercise (Experimental): 150 ug glucagon will be administered subcutaneously just before exercise
  Interventions: Drug: GlucaGen
- Control (No Intervention): No glucagon will be administered before exercise

INTERVENTIONS:
Drug: GlucaGen — 150 ug glucagon will be administered to the participants before exercise.
  Other Names: Glucagon, GlucaGen®, Novo Nordisk, ATC code H04AA01
  Arms: 150 ug glucagon before exercise

SUMMARY:
The primary aim of the study is to evaluate the glucose response to low-dose glucagon (single 150 µg dose) administered immediately before aerobic exercise in individuals with AHCL-treated T1D.

DETAILED DESCRIPTION:
The study consists of a screening visit (visit A) and two additional study visits (visit B and visit C) completed in a sequential order. During study visit B participants will receive s.c. administration of 150 ug glucagon prior to a 45-min moderate intensity continuous exercise session and subsequently continue into a 1-hour post-exercise observation period. During study visit C the exact same procedures will be followed with the omission of glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type 1 diabetes ≥ 2 years
* Use of AHCL system MiniMed 780G ≥ 4 weeks
* Use of Novorapid for ≥ 1 week

Exclusion Criteria:

* Allergies to lactose or glucagon
* Known or suspected allergies to glucagon or related products
* History of hypersensitivity or allergic reaction to glucagon or lactose
* Patients with diagnosed pheochromocytoma, insulinoma or gastroparesis
* Concomitant medical or psychological conditions identified through review of medical history, physical examination and clinical laboratory analysis that, according to the investigator's assessment, makes the individual unsuitable for study participation
* Lack of compliance with key study procedures at the discretion of the investigator
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (methods are considered adequate for study enrolment for females: an intrauterine device, hormonal contraception (birth control pills, implant, patch, vaginal ring or injection), a single partner who is sterile or infertile, or sexual abstinence. Contraception is required throughout the study duration. Sterilized or postmenopausal women (>12 months since last period) are not required to use contraception)
* Inability to understand the individual information and to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sissel B Lundemose, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross-over study. A total of 10 unique participants were enrolled and assigned to both arms sequentially. Therefore, the number of participants started in each arm is 10, but these represent the same individuals.
  We initially planned for 16 participants, but only 10 participants completed both visits.
Period: Visit B
Arm/Group | 150 ug Glucagon Before Exercise | Control
Started | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0
Period: Visit C
Arm/Group | 150 ug Glucagon Before Exercise | Control
Started | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 150 µg Glucagon Before Exercise Then No Glucagon Administered Before Exercise: All participants received 150 µg Glucagon before exercise during Visit B, followed by a control condition (no glucagon) during Visit C in a fixed sequence
Arm/Group | 150 µg Glucagon Before Exercise Then No Glucagon Administered Before Exercise
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 50 [42 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 10

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Time in Target Glucose Range (PG: 3.9 - 10.0 mmol/l) During and for 1-hour After Dynamic Physical Exercise Between Visit B and C
Description: This outcome measure evaluates the difference in the percentage of time participants spend within a specified glucose target range over a defined monitoring period. The measure aims to assess improvements or changes in glycemic control resulting from the intervention under study.
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: Percentage of time in range
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
Percentage of time in range | 100 [91 to 100] | 100 [100 to 100]

2. Secondary Outcome: Difference in Incidence Rate of Hypoglycaemic Events (PG<3.9 mmol/l) Between Visit B and C
Description: This outcome measure assesses the frequency of hypoglycemic events experienced by participants over a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Count of Participants; unit: Participants
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

3. Secondary Outcome: Difference in Time (Min) to Hypoglycaemia (PG<3.9 mmol/l) Between Visit B and C
Description: This outcome measure evaluates the time (in minutes) taken to reach hypoglycemia during a specified monitoring period or following a specific intervention.
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: minutes
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
minutes | NA [NA to NA] — Since no events of hypoglycaemia occured, this endpoint was not calculated. | NA [NA to NA] — Since no events of hypoglycaemia occured, this endpoint was not calculated.

4. Secondary Outcome: Difference in Percentage of Time Below Target Glucose Range (PG<3.9 mmol/l) Between Visit B and C
Description: as for outcome 1
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: percentage of time below range
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
percentage of time below range | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Difference in Percentage of Time Above Target Glucose Range (PG>10.0 mmol/l) Between Visit B and C
Description: as for outcome 1
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: percentage of time above range
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
percentage of time above range | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Difference in Incidence Rate of Hyperglycaemia (PG>10.0 mmol/l) Between Visit B and C
Description: This outcome measure assesses the incidence rate of hyperglycemia during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Number; unit: participants
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
participants | 0 | 0

7. Secondary Outcome: Difference in Nadir PG Concentration Between Visit B and C
Description: This outcome measure assesses the difference in the lowest value of plasma glucose during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: mmol/l
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
mmol/l | 5.8 [5.2 to 6.9] | 5.8 [4.9 to 6.5]

8. Secondary Outcome: Difference in Peak PG Concentration Between Visit B and C
Description: This outcome measure assesses the difference in peak plasma glucose during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
mmol/l | 9.3 (1.8) | 7.5 (1.4)

9. Secondary Outcome: Difference in Incremental Peak PG Concentration Between Visit B and C
Description: This outcome measure assesses the difference in incremental peak of plasma glucose during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: mmol/l
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
mmol/l | 1.8 [0.9 to 2.3] | -0.6 [-0.8 to 0.1]

10. Secondary Outcome: Difference in Mean PG Concentration Between Visit B and C
Description: This outcome measure assesses the difference in mean plasma glucose during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
mmol/l | 8.3 (1.8) | 6.7 (1.3)

11. Secondary Outcome: Difference in PG Area Under the Curve (AUC) Between Visit B and C
Description: This outcome measure assesses the difference in plasma glucose AUC during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: mmol/l*min
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
mmol/l*min | 824.2 [782.3 to 941.2] | 686.2 [612.6 to 821.1]

12. Secondary Outcome: Difference in Standard Deviation in PG Concentrations Between Visit B and C
Description: This outcome measure assesses the difference in SD plasma glucose during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Median (Full Range); unit: mmol/l
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
mmol/l | 1.0 [0.7 to 1.2] | 0.5 [0.3 to 0.6]

13. Secondary Outcome: Difference in Coefficient of Variation in PG Concentrations Between Visit B and C
Description: This outcome measure assesses the difference in CV in plasma glucose during a specified monitoring period.
Time Frame: 0 min to +105 min
Measure: Mean (Standard Deviation); unit: Percentage of variation
Arm/Group | 150 ug Glucagon Before Exercise | Control
Number analyzed (Participants) | 10 | 10
Percentage of variation | 12.3 (4.3) | 7.3 (2.5)

ADVERSE EVENTS:
Time Frame: Fromtime 0 until time 105, the entire trial.
Description: Visuel analouge scale (VAS) score 1-100
Arm/Group | 150 ug Glucagon Before Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT05379686/Prot_SAP_000.pdf